CLINICAL TRIAL: NCT01284686
Title: Pathophysiology of Neuronal Oscillations Within Subthalamo-cortical Loops in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2009-A00913-54
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Parkinson's Disease; Pathophysiology of Neuronal Oscillations Within Subthalamo-cortical Loops
Keywords: Pathophysiology; Parkinson; neuronal oscillations
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- dopamine (Active Comparator): ON DOPA:The patient will take his usual treatment with dopamine
  Interventions: Other: subthalamo-cortical loops stimulation in a one-sided and bipolar way
- without dopa (Experimental): OFF Dopa: The patient will be deprived of his treatment usual dopaminergique for at least 12 hours
  Interventions: Other: subthalamo-cortical loops stimulation in a one-sided and bipolar way

INTERVENTIONS:
Other: subthalamo-cortical loops stimulation in a one-sided and bipolar way — Record STN-cortex LFP coherence pattern and then stimulate STN (at 0, 5, 10, 15, 20, 25, 30 Hz) in newly implanted patients
  Arms: dopamine
Other: subthalamo-cortical loops stimulation in a one-sided and bipolar way — Record STN-cortex LFP coherence pattern and then stimulate STN (at 0, 5, 10, 15, 20, 25, 30 Hz) in newly implanted patients
  Arms: without dopa

SUMMARY:
Neuronal activity in circuits between the basal ganglia (BG) and motor cortical areas is abnormally synchronised and rhythmic. The oscillatory activity prevails at 8-30 Hz in untreated Parkinson's Disease (PD) and its amplitude at both subthalamic and cortical levels inversely correlates with motor impairment. Moreover, these different levels in BG-cortical loops are coherent in this frequency band. The 8-30 Hz activity is suppressed by treatment following treatment with dopaminergic drugs and is partially suppressed prior to and during voluntary movements. An unanswered question is how do BG-cortical loops become so prominently engaged in this oscillatory activity? One possible explanation is that the resonance frequencies of the loops fall in the 8-30 Hz band in the untreated state, so that oscillations in this band are transmitted particularly well. This hypothesis was confirmed in a previous series of experiments.The aim is to determine whether the resonance frequency within BG-cortical loops is correlated to the BG-cortical coherence frequency (with 20 subjets during 24 months).

DETAILED DESCRIPTION:
Methods: Record STN-cortex LFP coherence pattern and then stimulate STN (at 0, 5, 10, 15, 20, 25, 30 Hz) in newly implanted patients at rest and during simple and complex motor tasks while recording the steady state evoked potential over the cortex using EEG. The resonance frequency will be calculated as previously (Eusebio et al, Brain 2009). Experiments will be carried out both in the OFF medication and ON medication condition.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease idiopathique evolving for more than 5 years
* Dopa-Sensibility superior to 50 %
* Electrodes of stimulation implanted in 2 NST at Timone (Pr PERAGUT)

Exclusion Criteria:

* Bad tolerance of the condition OFF Dopa and\or OFF stimulation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-03-26 (Actual); Primary Completion 2015-05-27 (Actual); Study Completion 2015-05-27 (Actual)

PRIMARY OUTCOMES:
the understanding of the mechanisms underlying the propagation of pathological oscillatory activities in PD | 24 months

SECONDARY OUTCOMES:
may provide a basis for different therapeutic strategies | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe AZULAY, Principal Investigator — APHM
Locations (1):
- APHM, Marseille, France